CLINICAL TRIAL: NCT01917513
Title: Prospective Randomized Trial to Compare the Clinical Efficiency (Adenoma Detection Rate) of G-EYE™ HD Colonoscopy With Standard HD Colonoscopy
Brief Title: Prospective Trial to Compare the Clinical Efficiency of G-EYE™ HD Colonoscopy With Standard HD Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Smart Medical Systems Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: G-EYE 15505
Record Dates: First submitted 2013-07-30; First posted 2013-08-06 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2017-12

CONDITIONS: Adenoma; Polyps; Colorectal Cancer
Keywords: Adenoma; Polyps; CRC; Colonoscopy; Detection Yield
MeSH Terms: conditions — Adenoma; Polyps; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- G-EYE™ colonoscopy (Experimental): G-EYE™ colonoscopy
  Interventions: Device: G-EYE™ colonoscopy
- Standard Colonoscopy (Active Comparator): Standard Colonoscopy
  Interventions: Device: Standard Colonoscopy

INTERVENTIONS:
Device: G-EYE™ colonoscopy — G-EYE™ colonoscopy
  Arms: G-EYE™ colonoscopy
Device: Standard Colonoscopy — Standard Colonoscopy
  Arms: Standard Colonoscopy

SUMMARY:
The purpose of this study is to compare the adenoma detection rate of G-EYE™ high definition colonoscopy with that of standard high definition colonoscopy

DETAILED DESCRIPTION:
This is a multicenter, two-arm, randomized, open-label study intended to compare the detection rate obtained by performing G-EYE™ high definition colonoscopy vs. the detection rate obtained by performing high definition standard colonoscopy.

The study will enroll 1000 subjects. Consecutive adult subjects who were referred for elective colonoscopy will be asked to enroll into this randomized clinical study if the candidate meets the study inclusion and exclusion criteria.

Subjects will sign informed consent form and undergo randomization. The study includes a run-in preliminary phase of 270 patients to allow physicians to get familiar with the G-EYE™ endoscope.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 50 years old
2. Referred to colonoscopy for screening, following positive FOBT testing, change of bowel habits or for surveillance colonoscopy (history of adenoma resection).
3. The patient must understand and provide written consent for the procedure.

Exclusion Criteria:

1. Subjects with inflammatory bowel disease;
2. Subjects with a personal history of polyposis syndrome;
3. Subjects with suspected chronic stricture potentially precluding complete colonoscopy;
4. Subjects with diverticulitis or toxic megacolon;
5. Subjects with a history of radiation therapy to abdomen or pelvis;
6. Pregnant or lactating female subjects;
7. Subjects who are currently enrolled in another clinical investigation.
8. Subjects with current oral or parenteral use of anticoagulants
9. Subjects with recent (within the last 3 mounts) coronary ischemia or CVA (stroke)
10. Any patient condition deemed too risky for the study by the investigator
11. Previous colonic surgery (except for appendectomy)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Kiesslich, Prof., Principal Investigator — Helios Dr. Horst Schmidt Kliniken, Wiesbaden, Germany
Locations (15):
- United States (2):
  - Beth Israel Deaconess Medical Center, Harvard Medical School, Boston, Massachusetts
  - NYU Langone Medical Center, New York, New York
- Herlev Hospital, Harlev, Denmark
- Germany (3):
  - Universitätsmedizin Johannes Gutenberg University Mainz, Mainz
  - Universitätsklinikum Tübingen, Tübingen
  - Helios Dr. Horst Schmidt Kliniken (HSK), Wiesbaden
- Asian Institute of Gastroenterology, Hyderabad, India
- Israel (3):
  - Hadassah Medical Center, Jerusalem
  - Laniado Hospital, Netanya
  - Assaf Harofeh Medical Center, Tzrifin
- Vita Salute San Raffaele University - Scientific Institute San Raffaele, Milan, Italy
- Netherlands (2):
  - Maastricht University Medical Centre, Maastricht
  - Radboud UMC, Nijmegen
- United Kingdom (2):
  - Birmingham City University, Birmingham
  - Russells Hall Hospital, Dudley

REFERENCES:
- [Derived] Shirin H, Shpak B, Epshtein J, Karstensen JG, Hoffman A, de Ridder R, Testoni PA, Ishaq S, Reddy DN, Gross SA, Neumann H, Goetz M, Abramowich D, Moshkowitz M, Mizrahi M, Vilmann P, Rey JW, Sanduleanu-Dascalescu S, Viale E, Chaudhari H, Pochapin MB, Yair M, Shnell M, Yaari S, Hendel JW, Teubner D, Bogie RMM, Notaristefano C, Simantov R, Gluck N, Israeli E, Stigaard T, Matalon S, Vilkin A, Benson A, Sloth S, Maliar A, Waizbard A, Jacob H, Thielsen P, Shachar E, Rochberger S, Hershcovici T, Plougmann JI, Braverman M, Tsvang E, Abedi AA, Brachman Y, Siersema PD, Kiesslich R. G-EYE colonoscopy is superior to standard colonoscopy for increasing adenoma detection rate: an international randomized controlled trial (with videos). Gastrointest Endosc. 2019 Mar;89(3):545-553. doi: 10.1016/j.gie.2018.09.028. Epub 2018 Sep 28. PMID 30273591

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Colonoscopy: Patients in this group underwent standard high definition colonoscopy
- G-EYE™ Colonoscopy: Patients in this group underwent G-EYE™ high definition colonoscopy using using an insufflated balloon during withdrawal
Period: Overall Study
Arm/Group | Standard Colonoscopy | G-EYE™ Colonoscopy
Started | 502 | 498
Completed | 407 | 396
Not Completed | 95 | 102

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Colonoscopy | G-EYE™ Colonoscopy | Total
Number analyzed (Participants) | 396 | 407 | 803
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (8.79) | 65.4 (8.92) | 65.3 (8.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 173 | 204 | 377
  Male | 223 | 203 | 426

OUTCOME MEASURES:

1. Primary Outcome: Detection Rate of Adenomas and Serrated Lesions
Description: The percentage of patients with at least one adenoma or serrated lesion in the G-EYE™ group will be compared to the Standard group
Time Frame: Approximalty following 14 days (histology results)
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Colonoscopy | G-EYE™ Colonoscopy
Number analyzed (Participants) | 392 | 404
Participants | 147 | 194

2. Secondary Outcome: Number of Polyp and Adenoma Detection, Procedure Times and Safety (Number of Patients With Adverse Events.
Description: The secondary outcome is a composite-each of the measured parameters will be reported as a single value for each arm
Time Frame: Up to 14 days (histology results)
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | G-EYE™ Colonoscopy | Standard Colonoscopy
Serious Adverse Events (participants affected / at risk) | 2/502 | 0/498
Other Adverse Events (participants affected / at risk) | 0/502 | 0/498
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | G-EYE™ Colonoscopy (N=502) | Standard Colonoscopy (N=498)
obstructive sigmoid tumor (Gastrointestinal disorders) | 1 | 0
an irregular heart rate and bradycardia prior to the initiation of the procedure (Cardiac disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2013-07-09): https://cdn.clinicaltrials.gov/large-docs/13/NCT01917513/Prot_000.pdf